CLINICAL TRIAL: NCT02980406
Title: The Role of FODMAPs in Upper GI Effects, Colonic Motor Activity and Gut-brain Signaling at the Behavioral Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: FODMAP1
Record Dates: First submitted 2016-11-02; First posted 2016-12-02 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: FODMAP; Irritable bowel syndrome; Gastric accommodation; Gastric motility; brain-gut axis
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet; Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Fructans (Active Comparator): Fructans (FODMAP) are oligosaccharides containing fructose chains. Since the human body lacks hydrolases to break down these saccharides, fructans are poorly absorbed molecules in everybody. The fructan solution used in this study has a concentration of 38g/L.
  Interventions: Dietary Supplement: FODMAP
- Fructose (Active Comparator): Fructose can be found in the diet as free fructose, in sucrose or as polymer structure in fructans. Absorption varies and occurs more rapidly in the presence of glucose than for free fructose because glucose cotransport is involved in the uptake of fructose. Therefore, when fructose is in excess of glucose, it is regarded as a FODMAP. The fructose concentration used in this study is 100g/L.
  Interventions: Dietary Supplement: FODMAP
- FODMAP mix (Active Comparator): The FODMAP mix consists of 20g fructans, 10g galacto-oligosaccharides (GOS), 30g fructose, 10g sorbitol and 10g mannitol in one liter of tap water.
  Interventions: Dietary Supplement: FODMAP
- Glucose (Placebo Comparator): Glucose is a carbohydrate that is not classified as FODMAP, and is therefore used as a control in this study. The concentration of the glucose solution in this study is 100g/L.
  Interventions: Dietary Supplement: Glucose (control)

INTERVENTIONS:
Dietary Supplement: FODMAP — Fermentable oligo-, di- and monosaccharides and polyols are poorly absorbed carbohydrates that are known to cause symptoms in IBS patients.
  Arms: FODMAP mix; Fructans; Fructose
Dietary Supplement: Glucose (control) — Glucose is not a FODMAP.
  Arms: Glucose

SUMMARY:
In this study, the investigators aim to assess the effect of acute FODMAP infusion on gastric motility and on gastrointestinal and psychological symptoms. 20 healthy volunteers and 20 patients with irritable bowel syndrome (IBS) will undergo respectively four and two/three pressure measurements of the stomach after an overnight fast as a measure for gastric motility. During this pressure measurement, which takes approximately 4 hours, one of four FODMAP or control solutions will be administered directly into the stomach through a nasogastric tube. Administration will be stopped when the participant is fully satiated. The four solutions that will be tested in healthy volunteers are (1) a fructan solution, (2) a fructose solution, (3) a FODMAP mix and (4) a glucose solution as a control. In IBS patients, only the fructan and glucose solution will be tested, where after they can choose to come for a third visit to test the fructose solution. The solutions will be tested on separate occasions in a randomized order.

During the pressure measurement, participants will be asked to complete several questionnaires: (1) a gastrointestinal symptom questionnaire to assess their gastrointestinal symptoms, (2) a satiation questionnaire during infusion of one of the solutions, (3) psychological questionnaires (POMS, SAM, PANAS and STAI) to evaluate possible psychological effects of FODMAP infusion.

The investigators hypothesize that there will be differences in gastric motility between healthy volunteers and IBS patients. Furthermore, it is hypothesized that gastrointestinal symptoms will be increased in IBS patients, and that FODMAP infusion will have more psychological effects in patients than in healthy volunteers.

DETAILED DESCRIPTION:
In this study, the investigators aim to assess the effect of acute FODMAP infusion on gastric motility and on gastrointestinal and psychological symptoms. This is a randomised, single-blinded, crossover study of different solutions, differing in FODMAP content. The four solutions that will be tested in healthy volunteers are (1) a fructan solution, (2) a fructose solution, (3) a FODMAP mix and (4) a glucose solution as a control. In IBS patients, only the fructan and glucose solution will be tested, where after they can choose to come for a third visit to test the fructose solution. The different solutions will be tested on separate occasions, three days to one week apart, in a randomised order.

The preparation of each study visit will be identical. After an overnight fast, participants will be asked to come to the clinic. To ensure a low baseline symptom level and low microbial gut activity, a diet low in fibre and fermentable carbohydrates will be followed the day prior to each test (information will be provided to assist this). Participants will be asked to refrain from alcohol, tea and coffee, and intense physical activity for at least 12 hours before participation. They will also be asked to refrain from smoking cigarettes at least one hour before the start of the experiment.

A high resolution manometry probe will be inserted through the nose into the stomach of the participant to assess intragastric pressure as a measure of gastric motility and gastric accommodation. In addition, an infusion tube will be positioned in the proximal stomach to administer the solution. The position of the probes will be checked fluoroscopically (maximum 15 seconds). In this case, relevant guidelines of radioprotection will be adhered to. Patients will be protected by a lead shield that covers the lower abdomen and all personnel will wear a lead jacket. After the catheters are fixed to the subjects' chin, the patients will be asked to sit at a table and remain in this position for the remainder of the experiment.

After a stabilization period of at least 15 minutes, and when the subject is in phase II of the hunger cycle, one of four solutions will be intragastrically administered at a constant speed of 60 mL per minute (determined by an automated system using a peristaltic pump). IGP will be recorded for the duration of the drink infusion and for the following 3 hours. During infusion, the subjects will be asked to score their satiation at 1-minute intervals using a graphic rating scale that combines verbal descriptors on a scale graded of 0-5 (1, threshold; 5, maximum satiety). The intragastric infusion will be stopped as soon as a score of 5 is reached on their satiation scores. In addition, participants will be asked to complete a gastrointestinal symptom questionnaire every 15 minutes. The participant's emotions and mood will be assessed before, immediately after and 1, 2 and 3 hours after infusion, using the State-Trait Anxiety Inventory (STAI) and the validated Dutch version of the Positive and Negative Affect Scale (PANAS). Emotional state will be repeatedly measured every 15 minutes using the Self-Assessment Manikin (SAM) and Profile of Mood States (POMS)-Fatigue subscale.

ELIGIBILITY:
Healthy volunteers:

Inclusion Criteria:

* Aged between 18 to 65 years old

Exclusion Criteria:

* Current symptoms or history of gastrointestinal disease, other significant diseases, psychological disorders, drug allergies or pregnancy
* Taking any medication or have any drug history

IBS patients:

Inclusion Criteria:

* Meet Rome III criteria for IBS. This is defined as recurrent abdominal pain or discomfort at least 3 days/month in the last 3 months associated with two or more of the following: improvement with defecation; onset associated with a change in frequency of stool; or onset associated with a change in form (appearance) of stool
* Aged between 18 to 65 years old

Exclusion criteria:

* Other significant diseases, psychological disorder, drug allergies or pregnancy
* Taking any non-steroidal anti-inflammatory drugs (NSAIDs), corticosteroids or other immunosuppressive drugs in the preceding 6 months. All drugs potentially affecting gastrointestinal motility or sensitivity will be discontinued at least 1 week before the gastric emptying study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in intragastric pressure measured by high resolution manometry | up to 3 hours after administration
  Intragastric pressure will be assessed as a measure for gastric accommodation and gastric motility

SECONDARY OUTCOMES:
Change in subjective gastrointestinal symptom scores measured by visual analogue scale of 100 mm | assessment by questionnaire (100 mm Visual Analogue Scale) every 15 minutes, up to 3 hours after administration
Change in mood/emotion measured by Profile Of Mood States (POMS) questionnaire. | POMS (Profile Of Mood States) every 15 minutes up to 3 hours after administration.
Change in mood/emotion measured by Self Assessment Manikin (SAM) questionnaire. | SAM (Self Assessment Manikin) every 15 minutes up to 3 hours after administration.
Change in mood/emotion measured by Positive and Negative Affect Scale (PANAS). | PANAS (Positive And Negative Affect Scale) before, after, 1h, 2h and 3h after administration.
Change in mood/emotion measured by State Trait Anxiety Index questionnaire. | STAI (State Trait Anxiety) before, after, 1h, 2h and 3h after administration.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, MD, PhD, Principal Investigator — UZ Leuven / KU Leuven

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Masuy I, Van Oudenhove L, Tack J, Biesiekierski JR. Effect of intragastric FODMAP infusion on upper gastrointestinal motility, gastrointestinal, and psychological symptoms in irritable bowel syndrome vs healthy controls. Neurogastroenterol Motil. 2018 Jan;30(1). doi: 10.1111/nmo.13167. Epub 2017 Aug 1. PMID 28762592